CLINICAL TRIAL: NCT04005261
Title: Is it Time to Revise Type 2 Diabetes Treatment: C-peptide Concentrations in Type 2 Diabetes Treated With Insulin
Brief Title: C-peptide Concentrations in Type 2 Diabetes Treated With Insulin; is it Time to Revise the Treatment of Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal Investigator, Goztepe Training and Research Hospital
Other Study IDs: C-peptide2019
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Type 2 diabetes; C-peptide; beta-cell reserve; insulin use
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with type 2 diabetes treated with insulin: Patients with type 2 diabetes who have been using insulin for at least six months.
  They should be older than 18 years The patients should be presented to the Diabetes Outpatient Clinics of Istanbul Medeniyet University Goztepe Training and Research Hospital
  Interventions: Diagnostic Test: C-peptide concentrations

INTERVENTIONS:
Diagnostic Test: C-peptide concentrations — The patients will be grouped by their C-peptide concentrations

SUMMARY:
C-peptide is used to evaluate beta cell reserves. Patients with type 2 diabetes are treated with insulin for different indications. Other than beta-cell insufficiency and organ failures, insulin treatment is needed for a specified period. The investigators want to evaluate beta cell reserves in patients with type 2 diabetes treated with insulin for at least six months to see if that is the case. The investigators also want to compare the characteristics of these patients according to their beta cell reserves.

DETAILED DESCRIPTION:
In patients with type 2 diabetes, initiation of insulin therapy is indicated in several conditions such as severe insulin resistance, acute metabolic decompensations, surgery, pregnancy, and progression of diabetic complications, and also when glycemic control cannot be achieved with effective lifestyle regulation and non-insulin antidiabetic medications. Some of these indications are transient, and patients should be reassessed to choose the appropriate treatment options. Clinical inertia is one of the new topics expressed in the recent diabetes guidelines. The investigators aimed to investigate the beta cell reserves of the patients with type 2 diabetes who are treated with insulin, to see if they have insufficient insulin secretion and if not, to compare their characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes who had been treated with insulin as a monotherapy or as a component of combination therapy for at least 6 months.

Exclusion Criteria:

* Diagnosis of other types of diabetes,
* end-stage renal failure,
* history of renal transplantation,
* diabetic acute metabolic decompensation,
* decompensated heart failure,
* advanced liver disease,
* pregnancy,
* acute or chronic pancreatitis,
* pancreatic carcinoma,
* acute infections,
* use of medications that might affect glucose regulation (e.g. corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with type 2 diabetes treated with insulin aged 18 years or older who presented to the Diabetes Outpatient Clinics of Istanbul Medeniyet University Goztepe Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adequate, borderline and insufficient beta cell reserves assessed by the fasting C-peptide concentrations | 3 months
  Fasting C-peptide concentrations will be measured in patients with type 2 diabetic patients using insulin as a monotherapy or as part of combination therapy and the patients will be grouped as patients with adequate beta cell reserves, patients with borderline beta cell reserves and patient with insufficient beta cell reserves.
Correlations of fasting C-peptide concentrations with patients characteristics and biochemical findings | 3 months
  Correlations of fasting C-peptide concentrations with patients characteristics and biochemical findings, especially the components of metabolic syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe N Erbakan, MD, Principal Investigator — IMU Doctoral program; Mehmet Uzunlulu, Prof, Study Director — IMU Goztepe Education and Research Hospital
Locations (1):
- IMU Goztepe Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leighton E, Sainsbury CA, Jones GC. A Practical Review of C-Peptide Testing in Diabetes. Diabetes Ther. 2017 Jun;8(3):475-487. doi: 10.1007/s13300-017-0265-4. Epub 2017 May 8. PMID 28484968
- [Background] Palmer JP, Fleming GA, Greenbaum CJ, Herold KC, Jansa LD, Kolb H, Lachin JM, Polonsky KS, Pozzilli P, Skyler JS, Steffes MW. C-peptide is the appropriate outcome measure for type 1 diabetes clinical trials to preserve beta-cell function: report of an ADA workshop, 21-22 October 2001. Diabetes. 2004 Jan;53(1):250-64. doi: 10.2337/diabetes.53.1.250. PMID 14693724
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S90-S102. doi: 10.2337/dc19-S009. PMID 30559235
- [Background] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, DeFronzo RA, Einhorn D, Fonseca VA, Garber JR, Garvey WT, Grunberger G, Handelsman Y, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez GE. CONSENSUS STATEMENT BY THE AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY ON THE COMPREHENSIVE TYPE 2 DIABETES MANAGEMENT ALGORITHM - 2019 EXECUTIVE SUMMARY. Endocr Pract. 2019 Jan;25(1):69-100. doi: 10.4158/CS-2018-0535. No abstract available. PMID 30742570
- [Result] Jones AG, Hattersley AT. The clinical utility of C-peptide measurement in the care of patients with diabetes. Diabet Med. 2013 Jul;30(7):803-17. doi: 10.1111/dme.12159. PMID 23413806
- [Derived] Uzunlulu M, Oguz A, Arslan Bahadir M, Erbakan AN, Vural Keskinler M, Alpaslan Mesci B. C-peptide concentrations in patients with type 2 diabetes treated with insulin. Diabetes Metab Syndr. 2019 Nov-Dec;13(6):3099-3104. doi: 10.1016/j.dsx.2019.11.010. Epub 2019 Nov 20. PMID 31785503